CLINICAL TRIAL: NCT06962813
Title: Transdermal Radiofrequency (V ERASER) Versus Polidocanol Sclerotherapy for the Treatment of Reticular Veins and Telangiectasias: A Randomized Controlled Trial (TYPER Trial)
Brief Title: Transdermal Radiofrequency V ERASER Versus Polidocanol Sclerotherapy for Reticular Veins and Telangiectasias
Acronym: TYPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Responsible Party: Principal Investigator, Eduardo Ramacciotti, Senior investigator, Science Valley Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYPER TRIAL
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Varicose Veins Leg; Telangiectasias
Keywords: radiofrequency; sclerotherapy; varicose veins
MeSH Terms: conditions — Telangiectasis; Varicose Veins

STUDY DESIGN:
Intervention Model Description: 2 arm parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency V Eraser (Experimental): radiofrequency
  Interventions: Procedure: Radiofrequency V Eraser
- Polidocanol sclerotherapy (Active Comparator): Standard of care, varicose veins, sclerotherapy
  Interventions: Procedure: Radiofrequency V Eraser

INTERVENTIONS:
Procedure: Radiofrequency V Eraser — standar of care sclerotherapy

SUMMARY:
This study tested V Eraser, Transdermal radiofrequency versus polidocanol sclerotherapy for the treatment of reticular veins and telangiectasia of the legs

DETAILED DESCRIPTION:
Chronic Venous Disease causes symptoms such as pain, edema, and skin manifestations, including telangiectasias and varicose veins. Sclerotherapy with polidocanol is the gold standard treatment; however, technologies such as laser devices and transdermal radiofrequency are also available. The V Eraser, a device that combines transdermal radiofrequency and sclerotherapy, was developed to treat these conditions.

Methods: This was a prospective, randomized, and comparative study comparing V Eraser with sclerotherapy for the treatment of telangiectasias and reticular veins. Forty-one patients were randomized to either V Eraser or polidocanol sclerotherapy and underwent a single treatment session. Efficacy was assessed using the Aberdeen Varicose Vein Questionnaire and vessel clearance analysis in pre- and post-treatment images.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign informed consent
* Patients from 18 to 80 years old with CVD classified as CEAP clinical classes C1 to C5, but only telangiectasias and reticular veins not connected to larger varicosities

Exclusion Criteria:

* Patients with great saphenous or small saphenous vein insufficiency.
* Patients with allergies to polidocanol
* Patients with contraindications to treat varicose veins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Photographic analysis | 30 days
  Image analysis of photos was performed on day 30. Using the ImageJ software, two blinded evaluators analyzed the pre- and post-procedure photographs, measuring the vessel lengths in both images
Aberdeen AVVQ questionnaire | 30 days
  The Aberdeen Varicose Vein Questionnaire (AVVQ) was applied on day 30

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca Higino, MD, Principal Investigator — Faculty of Medical Sciences of Santa Casa de São Paulo
Locations (1):
- Hospital São Luiz Gonzaga and Hospital da Irmandade Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno-Moraga J, Pascu ML, Alcolea JM, Smarandache A, Royo J, David F, Trelles MA. Effects of 1064-nm Nd:YAG long-pulse laser on polidocanol microfoam injected for varicose vein treatment: a controlled observational study of 404 legs, after 5-year-long treatment. Lasers Med Sci. 2019 Sep;34(7):1325-1332. doi: 10.1007/s10103-019-02736-1. Epub 2019 Feb 1. PMID 30707327
- [Background] Siribumrungwong B, Noorit P, Reanpang T, Pornwaragorn C, Wilasrusmee C, Wongsuwanich S, Srikuea K, Orrapin S, Benyakorn T, Garratt AM, Rerkaserm K. Reliability, validity, and minimal clinically important differences for the Thai-version of the Aberdeen Varicose Vein Questionnaire (AVVQ-Thai) in patients with chronic venous disease. F1000Res. 2024 Oct 11;13:486. doi: 10.12688/f1000research.147716.2. eCollection 2024. PMID 39925999
- [Background] Diken AI, Alemdaroglu U, Ozyalcin S, Hafez I, Tunel HA, Yalcinkaya A, Ecevit AN. Adjuvant radiofrequency thermocoagulation improves the outcome of liquid sclerotherapy in the treatment of spider veins of the leg: A pilot study. Phlebology. 2021 Sep;36(8):620-626. doi: 10.1177/02683555211006534. Epub 2021 Apr 4. PMID 33813962
- [Background] Key DJ. A Preliminary Study of a Transdermal Radiofrequency Device for Body Slimming. J Drugs Dermatol. 2015 Nov;14(11):1272-8. PMID 26580877
- [Background] Gloviczki P, Lawrence PF, Wasan SM, Meissner MH, Almeida J, Brown KR, Bush RL, Di Iorio M, Fish J, Fukaya E, Gloviczki ML, Hingorani A, Jayaraj A, Kolluri R, Murad MH, Obi AT, Ozsvath KJ, Singh MJ, Vayuvegula S, Welch HJ. The 2022 Society for Vascular Surgery, American Venous Forum, and American Vein and Lymphatic Society clinical practice guidelines for the management of varicose veins of the lower extremities. Part I. Duplex Scanning and Treatment of Superficial Truncal Reflux: Endorsed by the Society for Vascular Medicine and the International Union of Phlebology. J Vasc Surg Venous Lymphat Disord. 2023 Mar;11(2):231-261.e6. doi: 10.1016/j.jvsv.2022.09.004. Epub 2022 Oct 12. PMID 36326210